CLINICAL TRIAL: NCT01915563
Title: Phase 2 Study of 60-min Rest After Successful Spontaneous Breathing Trial Before Extubation as a Tool for Reduction Post-extubation Failure.
Brief Title: Rest After Spontaneous Breathing Trial for Prevention of Post-extubation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Rafael Fernandez, Head of Critical Care Department, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBT Spain 001
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: Weaning Failure
Keywords: Mechanical ventilation; Weaning; Extubation failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBT and extubation (No Intervention): After a SBT patients will be extubated as usual
- SBT and rest 60 min before extubation (Experimental): After SBT patients will be reconnected to mechanical ventilation during 60 min before extubation
  Interventions: Procedure: REST

INTERVENTIONS:
Procedure: REST — After a SBT patients will be extubated as usual or reconnected to mechanical ventilation for 60 min before extubation.
  Arms: SBT and rest 60 min before extubation

SUMMARY:
To evaluate if a rest period before extubation after a successful SBT trial could reduce the extubation failure rate.

DETAILED DESCRIPTION:
Intubation and mechanical ventilation are related with several complications. This increased the risk of mortality of intensive care patients. So, we always look for an early extubation when patients are recovered for the trigger disease. In spite of standardized manoeuvres to decided readiness for extubation these are not quite good because it has been described a failure extubation rate of 5% and a reintubation rate of 15%. Furthermore several risk factors has been associated with a major failure rate:>65 years old, congestive cardiac insufficiency, chronic obstructive pulmonary disease, APACHE II >12 the extubation day, BMI >30, ineffective cough, a lot of bronchial secretions (as the need for >2 endotracheal suctioning in the last 8h before extubation), failure of a previous SBT,alterations of high respiratory tract or intubation for more than 7 days.Patients without any of these factors risk has an extubation failure rate of 10% while if any of these are present extubation failure increase to 30%.

The most used technique as a weaning trial is named spontaneous breathing trial (SBT). Some physiological aspects suggest that breathing through an endotracheal tube could be a really effort trial. So our hypothesis is that a period of rest after SBT and before extubation could reduce the extubation failure rate.

ELIGIBILITY:
Inclusion Criteria:

* patients ventilated for more than 12h and ready to perform a SBT

Exclusion Criteria:

* patients under 18 years old,
* tracheostomy,
* excessive bronchial secretions,
* agitation,
* hypercapnia during SBT and not resuscitation orders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernandez Rafael, MD, PhD, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa; Fernandez Maria del Mar, MD, PhD, Study Director — Hospital Universitari Mutua de Terrassa
Locations (1):
- Hospitales: Mutua de Terrassa,Médico-quirúrgico Jaen, Morales Messeguer, General de Albacete, Lorca, Málaga, Santiago, General de Catalunya, Joan XXIII Tarragona, La Fe-Valencia, Bellvitge, Moises Broggi, Mateu Orfila, Reina Sofia, Severo-Ochoa, Delfos, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez MM, Gonzalez-Castro A, Magret M, Bouza MT, Ibanez M, Garcia C, Balerdi B, Mas A, Arauzo V, Anon JM, Ruiz F, Ferreres J, Tomas R, Alabert M, Tizon AI, Altaba S, Llamas N, Fernandez R. Reconnection to mechanical ventilation for 1 h after a successful spontaneous breathing trial reduces reintubation in critically ill patients: a multicenter randomized controlled trial. Intensive Care Med. 2017 Nov;43(11):1660-1667. doi: 10.1007/s00134-017-4911-0. Epub 2017 Sep 22. PMID 28936675

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Slight number of patients were enrolled after reaching the planned sample due to information delay.
Period: Overall Study
Arm/Group | SBT and Extubation | SBT and Rest 60 Min Before Extubation
Started | 243 | 227
Completed | 243 | 227
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBT and Extubation | SBT and Rest 60 Min Before Extubation | Total
Number analyzed (Participants) | 243 | 227 | 470
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (15) | 65 (15) | 63.5 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Not registered | NA — Not registered | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Not registered | NA — Not registered | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  Spain | 243 | 227 | 470

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Extubation Failure
Description: Development of predefined criteria of respiratory insufficiency within 48 hours after scheduled extubation
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | SBT and Extubation | SBT and Rest 60 Min Before Extubation
Number analyzed (Participants) | 243 | 227
Participants | 58 | 24

2. Secondary Outcome: ICU Mortality
Time Frame: up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | SBT and Extubation | SBT and Rest 60 Min Before Extubation
Number analyzed (Participants) | 243 | 227
Participants | 12 | 10

ADVERSE EVENTS:
Arm/Group | SBT and Extubation | SBT and Rest 60 Min Before Extubation
Serious Adverse Events (participants affected / at risk) | 0/243 | 0/227
Other Adverse Events (participants affected / at risk) | 0/243 | 0/227

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No